CLINICAL TRIAL: NCT00834028
Title: Recurrence and Distant Metastases in Hepatocellular Carcinoma Treated by Transcatheter Arterial Chemoembolization : The Roles of VEGF, Cathepsin L, Endostatin, and Angiopoietin-2.
Brief Title: Recurrence and Distant Metastases in Hepatocellular Carcinoma Treated by Transcatheter Arterial Chemoembolization
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Zu-Yau Lin/Kaohsiung Medical University Hospital, Kaohsiung Medical University Hospital
Other Study IDs: KMUH-IRB-950168
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2006-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; vascular endothelial growth factor; angiopoietin; cathepsin
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: patients with hepatocellular carcinoma receive transcatheter arterial chemoembolization

SUMMARY:
This project will include at least 40 patients with hepatocellular carcinoma (HCC) who will receive transcatheter arterial chemoembolization (TACE) as a sole method for the management. The serum is collected before and at the 3rd and 7th day after TACE. The serum levels of vascular endothelial growth factor, angiopoietin 2, endostatin and cathepsin L are determined. All patients will be evaluated according to the TNM system for the cancer staging before and 3 months after each session of treatment. The vascularity of tumor, the drug and the dose used for embolization, and the area of infarction will be recorded. These data will be compared with the clinical courses of the patients to obtain the most suitable way in the management of these patients.

DETAILED DESCRIPTION:
Transcatheter arterial chemoembolization (TACE) is the traditional method for the palliative management of patients with hepatocellular carcinoma (HCC). This method will cause tissue hypoxia in area of embolization. Several proangiogenic factors will be induced by the condition of hypoxia. This may have the possibility to promote the proliferation of the residual cancer cells. However, there is no study to clarify this issue. This project will determine the serial changes of serum proangiogenic factors (vascular endothelial growth factor, angiopoietin 2), antiangiogenic factor (endostatin) and cathepsin L before and after TACE. These data will be compared with the clinical courses of the patients to obtain the most suitable way in the management of these patients.

This project will include at least 40 patients with HCC who will receive TACE as a sole method for the management. The serum is collected before and at the 3rd and 7th day after TACE. The serum levels of vascular endothelial growth factor, angiopoietin 2, endostatin and cathepsin L are determined. All patients will be evaluated according to the TNM system for the cancer staging before and 3 months after each session of treatment. The vascularity of tumor, the drug and the dose used for embolization, and the area of infarction will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients with hepatocellular carcinoma treated by transcatheter arterial chemoembolization

Exclusion Criteria:

* patients with hepatocellular carcinoma unable to be treated by transcatheter arterial chemoembolization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
tumor progression | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: zu y lin, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan